CLINICAL TRIAL: NCT06134037
Title: Effects of Aminophylline Bolus on Eleveld and Schnider TCI (Target Controlled Infusion) Concentrations at Start and End of Burst Suppression Occurence and on BIS (Bispectral Index) During the Induction Phase of Total Intravenous Anaesthesia With TCI
Brief Title: Effects of Aminophylline Bolus on TCI (Target Controlled Infusion) Concentrations at Burst Suppression Occurence
Acronym: TCI
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Federico Linassi, MD, University of Padova
Other Study IDs: TeoBurst
Record Dates: First submitted 2023-11-10; First posted 2023-11-18 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia Brain Monitoring
MeSH Terms: interventions — Aminophylline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aminophylline: Patients who received Aminophylline bolus (4 mg/kg) at Burst Suppression occurence during induction of general anesthesia conducted with Eleveld TCI model
  Interventions: Drug: Aminophylline
- Not Aminophylline: Patients who did not received Aminophylline bolus (4 mg/kg) at Burst Suppression occurence during induction of general anesthesia conducted with Eleveld TCI model

INTERVENTIONS:
Drug: Aminophylline — Patients will be observationally included in the Aminophylline or not Aminiophylline group depending on anesthesiologist's discretion.
  Groups: Aminophylline

SUMMARY:
Aminophylline is an intravenous drug commonly utilized for asthma. However, some preclinical studies and few case reports and case series have described its effects in lightining the anesthestic plan during Propofol anaesthesia with an intravenous bolus of 4 mg/kg.

Authors aimed to compare its effect during accidental episodes of Burst Suppression during the induction phase of total Intravenous Anaesthesia with Target Controlled Infusion (TIVA-TCI) routinely utilized for general anaesthesia in our hospital.

DETAILED DESCRIPTION:
Aminophylline is an intravenous drug commonly utilized for asthma. However, some preclinical studies and few case reports and case series have described its utility in decrease the timing of return of consciousness after Propofol anaesthesia with an intravenous bolus of 4 mg/kg, and also to lightining the anestetic plan (increase in Bipectral Index - BIS- values).

Authors aimed to compare its effect during accidental Burst Suppression episodes during the induction of total Intravenous Anasethesia with Target Controlled Infusion (TIVA-TCI) routinely utilized for general anaesthesia in our hospital, with Eleveld Pharmacokinetic/Pharmacodynamic-PK/PD model).

The timing and relative Concentration of Propofol (CeP) from the start to the end of Burst suppression episodes with or without aminophylline bolus deliveres as soon as detected were taken into account.

ELIGIBILITY:
Inclusion Criteria:

* Undergo general anaesthesia with Targeted Controlled Infusion of Propofol (Eleveld model) and Remifentanil (Minto model)
* Burst Suppression accidental occurence during the induction phase of anesthesia.

Exclusion Criteria:

* Neurological disease
* Psychiatric disease
* Obesity
* Hypothension during Burst Suppression episodes, other Burst suppression episodes during Anesthesia maintenance.

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women undergoing brast cancer surgery with general anesthesia with Propofol and Remifentanil TCI, with or without aminophylline bolus at Burst Suppression occurence during induction will be recruited
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-11-12 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Correlation between Concentration at the effector site of Propofol after Aminophylline bolus during Burst Suppression occurence | Authors will collected data about Drugs concentration and BIS values during general anaesthesia. We will collect BIS and TCI Propofol values during all the duration of anesthesia, form the start of anaesthesia until the emergence from anesthesia
  Discover if, after an aminophylline bolus, there are differences between Concentrations at the effector site of Propofol and timing of Burst Suppression duration during standard general anaesthesia conducted with Propofol and remifentanil delivered with target controlled infusion pumps, usually adopted in our Hospital to delivery general anaesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Treviso Regional Hospital, Treviso, TV, Italy